CLINICAL TRIAL: NCT04048239
Title: Development of a Robotic Minimally Invasive Pathway for Cochlear Implantation
Acronym: ROSA-IC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PI2019_843_0004
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Cochlear Hearing Loss; Implant
Keywords: cochlear implant; robotic; mini-invasive
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Cochlear Implantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cochlear implantation — cochlear implantation is a system developed to restore hearing in people with profound sensorineural hearing loss, whose classical hearing aids are ineffective. Surgery is necessary to insert the internal part into the cochlea and requires milling the mastoid to access the round window. This approach is technically difficult, and is performed under a microscope by an experienced surgeon.
Other: computerized tomography (CT) scan — computerized tomography (CT) scan of the facial nerve
Other: electromyograph — electromyographic verification of the facial nerve

SUMMARY:
Cochlear Implantation is a system developed to restore hearing in people with profound sensorineural hearing loss, whose classical hearing aids are ineffective. Surgery is necessary to insert the internal part into the cochlea and requires milling the mastoid to access the round window. This approach is technically difficult, and is performed under a microscope by an experienced surgeon. The development of a surgical technique that is both safer and less invasive is currently possible thanks to robotics.

DETAILED DESCRIPTION:
The ROSA robot coupled to the O-Arm scanner will guide the milling to the round window, whose path has been previously modeled, with the identification of the facial nerve. Milling will be done in 2 stages with a CT (computerised tomography scan) and electromyographic verification of the facial nerve. The insertion of the implant will be performed manually under endoscopic control. The preoperative and postoperative course of the patient will be identical.

ELIGIBILITY:
Inclusion Criteria:

* patients eligible for cochlear implantation in CHU Amiens
* patient more than 18 years old.

Exclusion Criteria:

* malformation or significant antecedent of mastoidectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
cochlear implantation with the ROSA robot surgery time | during surgery, day 1
  cochlear implantation with the ROSA robot surgery time
surgical quality based on material description and surgical technique | during surgery, day 1
  surgical quality based on material description and surgical technique

SECONDARY OUTCOMES:
surgical quality based on robot precision | during surgery, day 1
  surgical quality based on robot precision
surgical quality based on the cochlear implantation in the cochlea | during surgery, day 1
  surgical quality based on the cochlear implantation in the cochlea
surgical quality based on intraoperative electrophysiological data | during surgery, day 1
  surgical quality based on intraoperative electrophysiological data
surgical quality based on pathological complications | during surgery and postoperative period (1.5 month after surgery)
  surgical quality based on pathological complications (facial, paralysis, infection, pain)

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie klopp-Dutote, MD, Principal Investigator — CHU amiens
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Klopp-Dutote N, Lefranc M, Strunski V, Page C. Minimally invasive fully ROBOT-assisted cochlear implantation in humans: Preliminary results in five consecutive patients. Clin Otolaryngol. 2021 Nov;46(6):1326-1330. doi: 10.1111/coa.13840. Epub 2021 Aug 17. No abstract available. PMID 34310841